CLINICAL TRIAL: NCT07017478
Title: Mood Effects of Serotonin Agonists: Depression
Acronym: MESA-D
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IRB24-1947; 5R01DA002812-35 (NIH)
Record Dates: First submitted 2025-04-22; First posted 2025-06-12 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: LSD; Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): distilled water (0.26 mL)
  Interventions: Drug: Placebo
- LSD (26 micrograms) (Experimental): LSD tartrate in tasteless solution (0.26 mL)
  Interventions: Drug: LSD

INTERVENTIONS:
Drug: LSD — The serotonin 2A receptor agonist LSD
  Arms: LSD (26 micrograms)
Drug: Placebo — Distilled water
  Arms: placebo

SUMMARY:
This study will examine the effect of a low dose of the 5HT2A agonist LSD (26 µg), compared to placebo, on acute and protracted mood states in individuals with depression. The investigators will assess the relationship between mood-related symptoms and EEG as a neurophysiological marker.

DETAILED DESCRIPTION:
Depression is one of the leading mental health disorders in the U.S, with an estimated 21 million adults having at least one major depressive episode in the past year. Existing antidepressant medications have limited efficacy, undesirable side effects and can take weeks to months to provide relief of symptoms. Compounds that modulate serotonin 2A receptor signaling have potential to elicit rapid antidepressant effects, and one promising example of these compounds is lysergic acid diethylamide (LSD). There are widespread reports that very low doses of LSD improve mood and energy without producing hallucinogenic effects. Yet, these effects have not been rigorously tested under blinded, placebo-controlled conditions. There is an urgent need for controlled studies to assess the potential efficacy and the mechanisms that mediate any therapeutic effects.

In a preliminary double-blind, placebo-controlled study, the investigators found that depressed individuals reported acute mood enhancing effects after a single low dose of LSD, as well as improvements in anhedonia and sleep disturbance related symptoms, for as long as two days after the dose (preliminary data). The mechanisms underlying these effects are not known. While the acute mood enhancing effects may be due to direct actions of the drug at serotonin 2A receptors, animal models suggest that the sustained antidepressant-like effects of LSD are mediated by enhanced neural plasticity. In healthy humans, low doses of LSD produce sustained neurophysiological changes detected via EEG and on sleep measures, some of which may be related to antidepressant effects. In animal models, LSD produces long-lasting antidepressant-like responses as well as increased synaptic and dendritic growth in cortical regions days after drug exposure. Notably, these changes in structural plasticity are dependent on brain derived neurotrophic factor (BDNF), a protein that peaks after 24 hours in animal models.

In the current study the investigators will examine acute and delayed improvements in mood following a single low dose of LSD, in individuals with major depressive disorder (MDD). The investigators will examine the mechanisms underlying these antidepressant effects by assessing drug-induced neurophysiological changes using depression-sensitive behavioral tasks, EEG, and changes in sleep quality and architecture.

ELIGIBILITY:
Inclusion Criteria:

* English Fluency
* high school education or higher
* BMI between 19-30 kg/m2

Exclusion Criteria:

* individuals with a medical condition contraindicating study participation as determined by the study physician (e.g., liver disease, abnormal EKG, liver or cardiovascular disease)
* high blood pressure (>140/90)
* current suicidal ideation or suicide attempt in past 12 months
* past year severe substance use disorder
* personal or first-degree relative with history of psychosis
* currently taking any psychiatric medication (for conventional antidepressants must be off for ≥ 2 weeks)
* active panic disorder
* severe obsessive-compulsive disorder
* severe post-traumatic stress disorder
* women who are pregnant or planning to become pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Acute Mood Measures | Peak change (~2 hours post-drug) from pre-drug baseline
  Acute (Profile of Mood States scale ratings from 0-60).
Acute Mood Measures | Peak change (~2 hours post-drug) from pre-drug baseline
  Acute (Visual Analog Scale questionnaires, scale ratings from 0-100).
Delayed Mood Measures | Change from baseline (orientation) to 48-hour followup
  Delayed depressed mood measures (Beck Depression Inventory [score range: 0-63, higher scores greater symptoms severity] and Inventory of depression and anxiety symptoms [score range: 0-48, higher scores increased severity])
Effort expenditure for reward (EEFRT) Behavioral Task Performance | 2 hours post-drug administration
  Effort Expenditure for Reward Task
Sleep Quality | Change from baseline (pre-drug) to Night 0, 1, and 2 post-drug
  Electroencephalogram (EEG) power to assess time spent in Rapid Eye Movemeent [REM] and slow wave sleep
Sleep Quality | Change from baseline (pre-drug) to Night 0, 1, and 2 post-drug
  subjective measures of sleep function (Karolinska sleep log)

SECONDARY OUTCOMES:
Self-reported feelings of connection using Likert scale conversation questionnaires | Collected at the end of the session, 270 minutes post-drug administration
  ratings of connectedness
Natural Language Processing using large language model | during 45 minute conversation, occurring 150 min after drug administration
  Differences in speech content across drug conditions will be assessed using a sentiment analysis score
Facial expression analysis using HUMEAI software for positive and negative affect | during 45 minute conversation, occurring 150 min after drug administration
  Changes in emotional facial expressions during conversations across drug conditions (positive, negative affect)
Self-Esteem implicit association test | 2 hours post drug
  Changes in Self-esteem IAT scores across drug conditions

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Molla, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duan W, Cao D, Wang S, Cheng J. Serotonin 2A Receptor (5-HT2AR) Agonists: Psychedelics and Non-Hallucinogenic Analogues as Emerging Antidepressants. Chem Rev. 2024 Jan 10;124(1):124-163. doi: 10.1021/acs.chemrev.3c00375. Epub 2023 Nov 30. PMID 38033123
- [Background] Husain MI, Ledwos N, Fellows E, Baer J, Rosenblat JD, Blumberger DM, Mulsant BH, Castle DJ. Serotonergic psychedelics for depression: What do we know about neurobiological mechanisms of action? Front Psychiatry. 2023 Feb 10;13:1076459. doi: 10.3389/fpsyt.2022.1076459. eCollection 2022. PMID 36844032
- [Background] Ling S, Ceban F, Lui LMW, Lee Y, Teopiz KM, Rodrigues NB, Lipsitz O, Gill H, Subramaniapillai M, Mansur RB, Lin K, Ho R, Rosenblat JD, Castle D, McIntyre RS. Molecular Mechanisms of Psilocybin and Implications for the Treatment of Depression. CNS Drugs. 2022 Jan;36(1):17-30. doi: 10.1007/s40263-021-00877-y. Epub 2021 Nov 17. PMID 34791625
- [Background] Murphy RJ, Muthukumaraswamy S, de Wit H. Microdosing Psychedelics: Current Evidence From Controlled Studies. Biol Psychiatry Cogn Neurosci Neuroimaging. 2024 May;9(5):500-511. doi: 10.1016/j.bpsc.2024.01.002. Epub 2024 Jan 26. PMID 38280630
- [Background] Walsh CA, Gorfinkel L, Shmulewitz D, Stohl M, Hasin DS. Use of Lysergic Acid Diethylamide by Major Depression Status. JAMA Psychiatry. 2024 Jan 1;81(1):89-96. doi: 10.1001/jamapsychiatry.2023.3867. PMID 37819655
- [Background] Ly C, Greb AC, Cameron LP, Wong JM, Barragan EV, Wilson PC, Burbach KF, Soltanzadeh Zarandi S, Sood A, Paddy MR, Duim WC, Dennis MY, McAllister AK, Ori-McKenney KM, Gray JA, Olson DE. Psychedelics Promote Structural and Functional Neural Plasticity. Cell Rep. 2018 Jun 12;23(11):3170-3182. doi: 10.1016/j.celrep.2018.05.022. PMID 29898390
- [Background] Moliner R, Girych M, Brunello CA, Kovaleva V, Biojone C, Enkavi G, Antenucci L, Kot EF, Goncharuk SA, Kaurinkoski K, Kuutti M, Fred SM, Elsila LV, Sakson S, Cannarozzo C, Diniz CRAF, Seiffert N, Rubiolo A, Haapaniemi H, Meshi E, Nagaeva E, Ohman T, Rog T, Kankuri E, Vilar M, Varjosalo M, Korpi ER, Permi P, Mineev KS, Saarma M, Vattulainen I, Casarotto PC, Castren E. Psychedelics promote plasticity by directly binding to BDNF receptor TrkB. Nat Neurosci. 2023 Jun;26(6):1032-1041. doi: 10.1038/s41593-023-01316-5. Epub 2023 Jun 5. PMID 37280397
- [Background] Allen N, Jeremiah A, Murphy R, Sumner R, Forsyth A, Hoeh N, Menkes DB, Evans W, Muthukumaraswamy S, Sundram F, Roop P. LSD increases sleep duration the night after microdosing. Transl Psychiatry. 2024 Apr 15;14(1):191. doi: 10.1038/s41398-024-02900-4. PMID 38622150
- [Background] Hutten NRPW, Quaedflieg CWEM, Mason NL, Theunissen EL, Liechti ME, Duthaler U, Kuypers KPC, Bonnelle V, Feilding A, Ramaekers JG. Inter-individual variability in neural response to low doses of LSD. Transl Psychiatry. 2024 Jul 15;14(1):288. doi: 10.1038/s41398-024-03013-8. PMID 39009578
- [Background] Bershad AK, Schepers ST, Bremmer MP, Lee R, de Wit H. Acute Subjective and Behavioral Effects of Microdoses of Lysergic Acid Diethylamide in Healthy Human Volunteers. Biol Psychiatry. 2019 Nov 15;86(10):792-800. doi: 10.1016/j.biopsych.2019.05.019. Epub 2019 Jun 3. PMID 31331617
- See also: Husain et al., 2022 — https://doi.org/10.3389/fpsyt.2022.1076459
- See also: Ling et al., 2022 — https://doi.org/10.1007/s40263-021-00877-y
- See also: Murphy et al., 2024 — https://doi.org/10.1016/j.bpsc.2024.01.002
- See also: Ly et al., 2018 — https://doi.org/10.1016/j.celrep.2018.05.022
- See also: Moliner et al., 2023 — https://doi.org/10.1038/s41593-023-01316-5
- See also: Allen et al., 2024 — https://doi.org/10.1038/s41398-024-02900-4
- See also: Hutten et al., 2024 — https://doi.org/10.1038/s41398-024-03013-8
- See also: Bershad et al., 2019 — https://doi.org/10.1016/j.biopsych.2019.05.019